CLINICAL TRIAL: NCT01438567
Title: A Randomised, Double-blind, Double-dummy, Parallel-group Multicenter Study to Demonstrate Improvement in Symptoms of Constipation and Non-inferiority in Analgesic Efficacy in Subjects With Non-malignant or Malignant Pain That Require Around-the-clock Opioid Therapy Taking 50/25 - 80/40 mg Twice Daily as Oxycodone/Naloxone Prolonged Release (OXN PR) Tablets Compared to Subjects Taking 50 - 80 mg Twice Daily Oxycodone Prolonged Release (OxyPR) Tablets Alone
Brief Title: A Study to Demonstrate Improvement in Symptoms of Constipation in Subjects That Require Around-the-clock Opioid Pain Killer Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OXN3506; 2010-021995-27
Record Dates: First submitted 2011-08-18; First posted 2011-09-22 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Pain; Constipation
Keywords: oxycodone naloxone combination; severe chronic and non-malignant pain; Malignant and non-malignant pain that requires around-the clock opioid therapy; Opioid related constipation
MeSH Terms: conditions — Pain; Constipation; Bronchiolitis Obliterans Syndrome | interventions — Oxycodone; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- OXN PR tablets (Experimental)
  Interventions: Drug: oxycodone/naloxone prolonged release (OXN PR) tablets
- OxyPR tablets (Active Comparator)
  Interventions: Drug: oxycodone prolonged release (OxyPR) tablets

INTERVENTIONS:
Drug: oxycodone/naloxone prolonged release (OXN PR) tablets — Drug: Oxycodone/naloxone prolonged release tablets Arms: OXN PR Dosage: 2x50/25mg daily or 2x60/30mg daily or 2x70/35mg daily or 2x80/40mg daily
  Arms: OXN PR tablets
Drug: oxycodone prolonged release (OxyPR) tablets — Drug: Oxycodone prolonged release tablets Arms: OxyPR Dosage: 2x50mg daily or 2x60mg daily or 2x70mg daily or 2x80mg daily
  Arms: OxyPR tablets

SUMMARY:
The primary research objective is to demonstrate that subjects taking OXN PR have improvement in symptoms of constipation as measured by the Bowel Function Index (BFI) compared to subjects taking OxyPR tablets alone with cancer and non-cancer related pain without reducing the effectiveness of pain relief as measured by the Brief Pain Inventory (BPI).

DETAILED DESCRIPTION:
The study OXN3506 is a multicentre, multiple-dose, randomised, double-blind, double-dummy, active-controlled, parallel-group study in male and female subjects with non-malignant or malignant pain requiring opioids to assess analgesic efficacy and symptoms of constipation secondary to opioid treatment. Subjects will be randomised to two treatment groups and will be treated with OXN PR or OxyPR for up to 5 weeks. The study is composed of three phases, a pre-randomisation phase, a double-blind phase and an extension phase.

ELIGIBILITY:
Inclusion Criteria

* Subjects who are receiving WHO step III opioid analgesic medication for the treatment of non-malignant or malignant pain.
* Documented history of non-malignant or malignant pain that requires around-the-clock opioid therapy

Exclusion Criteria

* Females who are pregnant or lactating.
* Subjects with evidence or significant structural abnormalities of the gastrointestinal tract.
* Subjects with evidence of impaired liver/kidney function upon entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Bowel function Index (BFI) | 5 weeks and a 6 month extension
  To demonstrate that subjects taking OXN PR have improvement in symptoms of constipation as measured by the Bowel Function Index (BFI) compared to subjects taking OxyPR

SECONDARY OUTCOMES:
Pain Intensity Scale (PIS) | 5 weeks
  To demonstrate non-inferiority of OXN PR compared to OxyPR with respect to the analgesic efficacy based on the subjects' 'Average Pain over last 24 Hours' assessed at each Double-blind Phase visit as measured by the Pain Intensity Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Ballygomartin Group Practice, Belfast, United Kingdom

REFERENCES:
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=OXN3506